

# Clinical Development

## CPPY988A1

# CPPY988A12201 (GT005-03) / NCT04566445

HORIZON: A Phase II, Open-Label, Outcomes-Assessor Masked, Multicenter, Randomized, Controlled Study to Evaluate the Safety and Efficacy of Two Doses of GT005 Administered as A Single Subretinal Injection in Subjects With Geographic Atrophy Secondary to Dry Age-Related Macular Degeneration

# **Statistical Analysis Plan (SAP)**

Document type: SAP Documentation

Document status: Amendment 3

Release date: 13-Jun-2024

Number of pages: 34

Property of Novartis
Confidential
May not be used, divulged, published or otherwise disclosed without the consent of Novartis

# Document History – Changes compared to previous final version of SAP Date Time Reason for Outcome for undate Section and to

| Date | Time<br>point | Reason for update | Outcome for update | Section and title impacted (Current) |
|---|---|---|---|---|
| 13-<br>July-<br>2023 | Prior<br>to<br>DB<br>lock | Creation of<br>final<br>version | N/A - First version | NA |
| 08- | Prior | • | Added Week 48 analysis and moved the | Section 1 |
| Jan-<br>2024 | to<br>DB<br>Lock | Amendment<br>1 | Week 72 analysis (primary objective) to the final analysis | Section 2.13 |
| | | | Revised the definition of estimand | Section 1.2.1 |
| | | | | Section 2.5 |
| | | | Updated the calculation of Study Day | Section 2.1.1 |
| | | | Removed the SAF | Section 2.2 |
| | | | Updated the analysis set used for patient disposition, demographics and other baseline characteristics | Section 2.3 |
| | | | Revised the analysis scope for prior, concomitant and post therapies | Section 2.4.2 |
| | | | Removed sensitivity and supplementary analyses for the primary objective | Section 2.5 |
| | | | Removed AEs by primary SOC, PT and maximum severity | Section 2.7.1 |
| | | | Added detailed information for PROs | Section 2.10 |
| | | | Added the analyses scope for Week 48 | Section 2.13 |
| | | | Revised the imputation rule | Section 5.1 |
| | | | Removed the analysis part for multiple imputation | Section 5.4 |

| Date | Time<br>point | Reason for update | Outcome for update | Section and title<br>impacted<br>(Current) |
|---|---|---|---|---|
| | | | | , |

# **Table of contents**

| | Table | of content | s | 4 |
|---|---|---|---|---|
| | List of | abbreviat | ions | 6 |
| 1 | Introdu | uction | | 7 |
| | 1.1 | Study de | esign | 7 |
| | 1.2 | Study ol | bjectives, endpoints and estimands | 9 |
| | | 1.2.1 | Primary estimand(s) | 11 |
| 2 | Statisti | ical metho | ods | 11 |
| | 2.1 | Data ana | alysis general information | 11 |
| | | 2.1.1 | General definitions | 12 |
| | 2.2 | Analysis | s sets | 13 |
| | | | | 13 |
| | 2.3 | Subject | disposition, demographics and other baseline characteristics | <del></del> 14 |
| | | 2.3.1 | Subject disposition | 14 |
| | | 2.3.2 | Demographics and other baseline characteristics | 14 |
| | | 2.3.3 | Medical history | 15 |
| | 2.4 | Treatme | ents (study treatment, rescue medication, concomitant therapies, compliance) | 15 |
| | | 2.4.1 | Study treatment | 15 |
| | | 2.4.2 | Prior, concomitant and post therapies | 16 |
| | 2.5 | Analysis | s supporting primary objective(s) | 16 |
| | | 2.5.1 | Primary endpoint(s) | 16 |
| | | 2.5.2 | Statistical hypothesis, model, and method of analysis | 16 |
| | | 2.5.3 | Handling of intercurrent events | 17 |
| | | 2.5.4 | Handling of missing values not related to intercurrent event | 17 |
| | | 2.5.5 | Sensitivity analyses | 17 |
| | | 2.5.6 | Supplementary analyses | 17 |
| | 2.6 | Analysis | s supporting secondary objectives | 17 |
| | | 2.6.1 | Secondary endpoint(s) | 18 |
| | | 2.6.2 | Statistical hypothesis, model, and method of analysis | 18 |
| | | 2.6.3 | Handling of missing values/censoring/discontinuations | 19 |
| | 2.7 | Safety a | nalyses | 19 |
| | | 2.7.1 | Adverse events (AEs) | 20 |
| | | 2.7.2 | Deaths | 21 |
| | | 2.7.3 | Loss in best corrected visual acuity | 21 |
| | | 2.7.4 | Laboratory data | 22 |
| | | 2.7.5 | Other safety data | 22 |
| | 2.8 | Pharmac | cokinetic endpoints | 23 |
| | 2.9 | PD and | PK/PD analyses | 23 |
| | 2.10 | Patient- | reported outcomes | 23 |

| | | | | 25 |
|---|-------|--------------|------------------------------------------|----|
| | | | | 25 |
| | 2.13 | Data ana | alysis at Week 48 | 27 |
| 3 | Samp | le size calc | culation | 28 |
| 4 | Chang | ge to proto | col specified analyses | 28 |
| 5 | Appe | ndix | | 29 |
| | 5.1 | Imputat | ion rules | 29 |
| | | 5.1.1 | AE date imputation | 29 |
| | | 5.1.2 | Concomitant medication date imputation | 31 |
| | 5.2 | AEs cod | ding/grading | 33 |
| | 5.3 | Laborate | ory parameters derivations | 33 |
| | 5.4 | Statistic | al models | 33 |
| | | 5.4.1 | Analysis supporting primary objective(s) | |
| | 5.5 | Rule of | exclusion criteria of analysis sets | 33 |
| 6 | Refer | ences | · | 34 |

# List of abbreviations

| List of abbre | eviations |
|---------------|------------------------------------------|
| AE | Adverse Event |
| AESI | Adverse Events of Special Interest |
| AMD | Age-related Macular Degeneration |
| ATC | Anatomical Therapeutic Chemical |
| BCVA | Best Corrected Visual Acuity |
| CFI | Complement factor I |
| CFP | Color Fundus Photography |
| CI | Confidence Interval |
| CIR | Copy Increment from Reference |
| CRO | Contract Research Organization |
| CSFT | Central Sub Field Thickness |
| CSR | Clinical Study Report |
| DBL | Database Lock |
| ETDRS | Early Treatment for Diabetic Retinopathy |
| FAF | Fundus autofluorescence |
| FAS | Full Analysis Set |
| FIR | Fist Interpretable Results |
| FRI | Functional Reading Independence |
| GA | Geographic atrophy |
| IOP | Intraocular Pressure |
| LLD | Low Luminance Difference |
| LLVA | Low-luminance Visual Acuity |
| LSM | Least-Squares Mean |
| MAR | Missing at Random |
| MMRM | mixed model repeated measures |
| MNRead | Minnesota low-vision Reading test |
| OCT | Optical Coherence Tomography |
| PD | Protocol Deviation |
| PT | Preferred Term |
| SAP | Statistical Analysis Plan |
| SD | Standard Deviation |
| SE | Standard Error |
| SOC | System Organ Class |
| TEAE | treatment-emergent Adverse Event |
| VFQ-25 | Visual Function Questionnaire-25 |
| WHO | World Health Organization |

#### 1 Introduction

The HORIZON study (CPPY988A12201) is being terminated early as Novartis has made the decision to stop the current clinical development program for GT005 in subjects with geographic atrophy (GA) based on the results from the futility interim analysis. All GT005-treated subjects will be transferred into the long-term safety follow-up study, ORACLE (CPPY988A12203B).

The purpose of this Statistical Analysis Plan (SAP) is to describe the implementation of the statistical analyses planned in/changed from the study protocol, and to provide detailed statistical methods that will be used for the HORIZON Clinical Study Report (CSR).

The analyses will be conducted at three time points as described below:

- The interim analysis for futility will be performed when approximately 60% of subjects have GA data available at Week 48
- The Week 48 analysis will be conducted when all enrolled subjects from both Stage 1 and Stage 2 complete (or discontinue prior to) the Week 48 Visit
- The final analysis will be conducted once all enrolled subjects complete (or discontinue prior to) the Week 96 visit and final Database Lock (DBL) is achieved

Details for the futility analysis will be described in a separate Data Monitoring Committee SAP. For the Week 48 analysis and the final analysis, data will be analyzed according to the data analysis plan described in this document that will be incorporated into the CSR.

A First Interpretable Results (FIR) document will be provided for the Week 48 analysis to document the corresponding analysis results based on the available data at the time of the analysis.

This SAP is based on the HORIZON Clinical Study Protocol V5.0, dated 15 September 2022.

## 1.1 Study design

This is a Phase II, open-label, outcomes-assessor masked, untreated-control, multicenter, randomized controlled study to evaluate the safety and efficacy of two doses of GT005 administered as a single-time subretinal injection in subjects with geographic atrophy (GA) secondary to dry age-related macular degeneration (AMD).

Approximately 250 subjects are planned to be randomized to one of two doses of GT005 or the untreated control group (2:1). Subjects who are screened, but not randomized, will be classed as Screen Failures and will be replaced.

Subjects entered the study must have genotyping and serum Complement factor I (CFI) evaluation performed by a Sponsor-approved laboratory, either through participation in another Gyroscope sponsored study or during the HORIZON screening period. Data from subjects screened in another Gyroscope sponsored study at the same investigative site as HORIZON may be used to fulfill the screening and eligibility requirements for this study. This is only permissible if the screening data is collected within the screening period specified in the clinical protocol. Following consent, subjects will undergo ophthalmic and clinical assessments to

determine eligibility for inclusion in the study. Should subjects fail to meet the eligibility for HORIZON, they will be classed as Screen Failures for this study and may be considered for entry into another Gyroscope sponsored study.

| On confirmation of eligibility, subjects will be randomized to one of two dose groups (medium dose, wg, or high dose, wg). Within each dose group, subjects will be allocated to GT005 or untreated control based on a 2:1 scheme. |
|---|
| Randomization/Stratification |
| Subjects will be randomized to medium dose vg), high dose vg), or untreate |
| control groups. |
| A permuted |
| block method will be used to obtain an approximately 2:1 ratio between the treatment grou and control within each dose group, within each stratum (Figure 1-1). |
| and control within each dose group, within each statum (11gure 11). |
| _ |
| _ |



The overall objective of the study is to evaluate safety and efficacy (anatomical and functional visual outcomes) of two doses of GT005 in subjects with GA due to AMD.

The primary efficacy endpoint of change from baseline in GA area at Week 72 will be assessed in the final analysis (Section 1) once the final DBL is achieved.





# 1.2 Study objectives, endpoints and estimands

Table 1-1 Objectives and related endpoints

| OBJECTIVES | ENDPOINTS Endpoint(s) for primary objective(s) |
|---|---|
| Primary objective(s) | |
| <ul> <li>To demonstrate the effect of GT005<br/>vs untreated control on the<br/>progression of GA in subjects with<br/>GA due to AMD</li> </ul> | The change from baseline to Week 72 in GA area as measured by FAF |

# • To evaluate the effect of GT005 on the progression of GA in subjects with GA due to AMD

- The change from baseline through Week 96 in GA area as measured by FAF
- To evaluate the safety and tolerability of GT005
- Frequency of treatment emergent adverse event (TEAE) through Week 96
- To evaluate the effect of GT005 on retinal anatomical measures
- Change in retinal morphology on multimodal imaging through Week 96
- To evaluate the effect of GT005 on functional measures
- Change in best corrected visual acuity (BCVA)
   Score via the early treatment for diabetic retinopathy (ETDRS) chart through Week 96
- Change in low luminance difference (LLD) via the ETDRS chart through Week 96
- To evaluate the effect of GT005 on visual function
- Change in reading performance as assessed by Minnesota low-vision reading test (MNRead) chart through Week 96
- Change in functional reading independence (FRI) index through Week 96
- To evaluate the effect of GT005 on patient-reported outcomes
- Change in quality of life measured on the visual function questionnaire-25 (VFQ-25) through Week 96



# 1.2.1 Primary estimand(s)

The primary estimand will focus on the effect attributable to different doses of GT005 on GA lesion size change from baseline based on FAF at Week 72 in subjects who have not received alternative GA medications or therapies in the study eye.

The primary estimand is described by the following attributes:

- 1. **Population:** Subjects with GA secondary to AMD. Details on the target population are defined by the study inclusion and exclusion criteria
- 2. Variable: Change from baseline in GA lesion size (mm<sup>2</sup>) based on FAF at Week 72
- 3. **Treatment:** The randomized treatment (different doses) of the investigational therapy GT005 delivered through transvitreal subretinal injection
- 4. **Summary measure:** The treatment difference of the variable means between GT005 (any dose) and untreated control divided by the variable mean of untreated control, represented as % difference relative to untreated control



#### 2 Statistical methods

# 2.1 Data analysis general information

The analyses will be performed by the Contract Research Organization (CRO) using SAS 9.4.

Categorical data will be presented as frequencies and percentages. For continuous data, mean, standard deviation, median, minimum, and maximum will be presented. These summary statistics will be presented by treatment group unless otherwise specified. Where appropriate, point estimates and confidence intervals (CI) of treatment differences will be provided.

#### 2.1.1 General definitions

#### 2.1.1.1 Study treatment

The following treatment groups will be presented:

- Untreated control
- Medium dose GT005 (
- High dose GT005 (vg)

## 2.1.1.2 Baseline and post-Baseline

Baseline (Day 1) is defined as

- the day following randomization for subjects randomized to untreated control
- the day of successfully receiving GT005 administration for subjects randomized to GT005
- or the latest surgery date for subjects who were randomized to GT005 but failed to receive GT005 administration on the first attempt to surgery

The baseline value for efficacy and safety variables is the last available value (scheduled or unscheduled) collected prior to the date of *Baseline*, or on the date of *Baseline* but prior to the time of GT005 administration for GT005 treatment groups.

All data collected after the date of *Baseline* are defined as post-baseline. The *study day* for a baseline or post-baseline scheduled or unscheduled visit is defined as:

$$Study \ day = \begin{cases} \text{(Date of visit) - (Date of randomization)} & \text{Untreated} \\ \text{(Date of visit) - (Date of treatment administration)} + 1 & \text{GT005} \end{cases}$$
The *study day* for a scheduled or unscheduled visit before baseline is defined as

$$Study \ day = \begin{cases} \text{(Date of visit)- (Date of randomization)} - 1 & \text{Untreated} \\ \text{(Date of visit)} - \text{(Date of treatment administration)} & \text{GT005} \end{cases}$$

### 2.1.1.3 End of study mapping

The end of study date is the date when a subject completes or discontinues the study. For reporting data by visit in outputs, the end of study visit will be allocated to the actual (reported) visit number. If the end of study date is not on a scheduled visit, then the end of study visit will be allocated, based on study day, to the closest future scheduled study visit.

### 2.1.1.4 Unscheduled visits

For unscheduled visits, the analysis visits will be derived with windowing where appropriate (e.g., Visit  $3 \pm 3$  days) as per the protocol. For scheduled visits, the analysis visits will be the actual (reported) visit number.

Data collected at unscheduled visits will not be used in 'by-visit' tabulations, graphs or analyses unless it can be mapped to a missed scheduled visit with the window specified per the protocol. If multiple unscheduled visits are allocated to the same missed scheduled visit:

- The unscheduled visit closest to the missed scheduled visit will be used
- If there are multiple unscheduled visits with the same distance to the missed scheduled visit, the latest one will be used

For analyses showing abnormalities, data from unscheduled visits will be considered individually, without mapping to a main visit.

For analyses based on all post-baseline values such as averages over a given period summaries of maximum/minimum values, data collected at unscheduled visits will be included.

All data collected at unscheduled visits will be listed.

#### 2.1.1.5 Missing baseline and post-baseline data

Missing baseline data will not be imputed.

Observations with values 'not done', 'not evaluable', 'not applicable' will be treated as missing values.

In case of multiple entries for the same assessment are observed within one visit, the latest assessment value will be used.

#### 2.1.1.6 Alternative GA medications or therapies

Avacincaptad pegol (Izervay) and pegcetacoplan (Syfovre) via intravitreal injection are Food and Drug Administration approved treatments for GA and are permittable alternative GA treatments in this study.

### 2.2 Analysis sets

The **All-Enrolled Set** includes all patients who signed informed consent. This analysis set will be used to summarize patient disposition.

The **Full Analysis Set (FAS)** will include all subjects who are randomized to GT005 or untreated control. The FAS will be used for the analysis of efficacy and safety data.

The number and percentage of subjects within each of the above analysis sets will be summarized.



# 2.3 Subject disposition, demographics and other baseline characteristics

#### 2.3.1 Subject disposition

Subject disposition (up to Week 48/Week 96) will be summarized separately by treatment group and total for the All-Enrolled Set: the number and percentage of screen failures (including the primary reason for screen failure), subjects enrolled, randomized, randomized and treated with GT005, completed a particular study period (Week 48/Week 96), discontinued the study prior to or at Week 48/Week 96 (including the primary reason for premature study discontinuation). For subject disposition up to Week 48, the number and percentage of ongoing subjects will also be provided.

In addition, protocol deviations (PDs) will be summarized by the number and percentage of subjects with each deviation category for the FAS.

### 2.3.2 Demographics and other baseline characteristics

Demographic and baseline characteristics including age, sex, race, (self-reported and genetically defined) ethnicity, and AMD genetic subgroup will be summarized with descriptive

statistics or number and percentage of subjects as appropriate by treatment group and in total for the FAS.

Baseline ocular characteristics for the study eye will be summarized by treatment group and in total for the FAS. Ocular baseline characteristics include:

- Study eye selection (left eye OS or right eye OD)
- Best corrected visual acuity BCVA (in ETDRS letters)
- Low-luminance visual acuity (LLVA) (in ETDRS letters)
- Low luminance deficit (LLD) (BCVA LLVA in ETDRS letters)
- GA lesion area (mm<sup>2</sup>) as assessed by FAF
- GA contour (Unifocal, Multifocal, Cannot Grade) as assessed by FAF
- GA foveal involvement (Foveal, Non-foveal, Cannot Grade) as assessed by FAF and optical coherence tomography (OCT)
- Junctional zone pattern (Atypical, Banded, Diffuse, Focal, Cannot Grade) as assessed by FAF
- Presence of hard drusen (Yes, No, Cannot Grade) as assessed by color fundus photography (CFP)
- Presence of soft drusen (Yes, No, Cannot Grade) as assessed by CFP
- Presence of calcified drusen (Yes, No, Cannot Grade) as assessed by CFP
- Presence of cuticular drusen (Yes, No, Cannot Grade) as assessed by CFP
- Presence of subretinal hemorrhage (Yes, No, Cannot Grade) as assessed by CFP
- Presence of intraretinal hemorrhage (Yes, No, Cannot Grade) as assessed by CFP
- Presence of reticular pseudodrusen (Yes, No, Cannot Grade) as assessed by OCT
- Central subfield thickness (CSFT) (µm) as assessed by OCT
- Years since GA diagnosis

## 2.3.3 Medical history

Medical histories/current medical conditions will be listed by treatment arm, including the reported term/PT/SOC, laterality if applicable, start/end date, ongoing status (Yes, No) indicating whether the event is ongoing by the time of analysis, etc.

# 2.4 Treatments (study treatment, rescue medication, concomitant therapies, compliance)

# 2.4.1 Study treatment

The FAS will be used for the analyses below.

GT005 is administered as a single-time subretinal injection into the study eye of subjects randomized to one of the two GT005 doses. The surgical procedure for subretinal administration

of GT005 is based on a standardized methodology. It is conducted by an appropriately qualified Vitreoretinal Surgeon in an operating room under appropriate anesthesia. Subjects allocated to the untreated control will not receive any treatment.

Study treatment will be summarized by the number and percentage of subjects randomized, subjects underwent study surgery, subjects treated with GT005, subjects who did not complete the study surgery successfully (including the primary reason for preventing successful completion of surgery, related/unrelated to the surgery procedure). The number and percentage of subjects discontinued study prior to surgery (including the primary reason for discontinuation) will also be provided.

#### 2.4.2 Prior, concomitant and post therapies

Prior medications are defined as drugs taken and stopped prior to the date of randomization. Any medication given at least once between the date of randomization and the last study visit will be a concomitant medication, including those that were started pre-randomization and continued after randomization. Prior or concomitant medication will be identified based on recorded or imputed start and end dates of taking the medication.

Prior and concomitant medications will be coded according to the WHO Drug Reference List dictionary with Anatomical Therapeutic Classification (ACT) class and preferred term (PT).

Concurrent procedures will be summarized by treatment group and in total for ocular (study eye and fellow eye) and non-ocular events, presented with the number and percentage of patients by System Organ Class (SOC) and PT.

Prior medications and concomitant medications will be listed by treatment arm, including the reported name of medication/standardized medication name, indication, route of administration, laterality if applicable, start/end date, etc.

# 2.5 Analysis supporting primary objective(s)

The primary objective of this study is to demonstrate the effect of GT005 vs untreated control on the progression of GA in subjects with GA due to AMD. This will be evaluated by measuring the GA area over time using FAF.

#### 2.5.1 Primary endpoint(s)

The primary endpoint is the change from baseline to Week 72 in GA area as measured by FAF.

#### 2.5.2 Statistical hypothesis, model, and method of analysis

The primary endpoint will be estimated among treatment groups via least-squares means from a mixed model repeated measures (MMRM) analysis with missing at random assumption. The model will include the change from baseline in GA area measured by FAF as the dependent variable, baseline GA area as the covariate, assessment visit, treatment group, two interaction terms (assessment visit and treatment group, assessment visit and baseline GA area) as the fixed effect and subject as a random effect.

An unstructured within subject correlation structure will be used for the covariance matrix. If the unstructured covariance matrix results in a lack of convergence then other covariance structures will be investigated. Toeplitz, First Order Autoregressive AR(1), and Compound Symmetry will be applied, in the specified order, until the model converges.

The estimated least-squares mean (LSM) for the change in GA area, and treatment difference of each GT005 dose against untreated control, as well as the corresponding 90% confidence interval, will be summarized by visit and treatment group. A line plot for the estimated LSM with 90% CI by visit and treatment group will also be provided.

#### 2.5.3 Handling of intercurrent events

The underlying question for the primary estimand is: what is the effect attributable to different doses of GT005 on GA change on FAF at Week 72 in subjects who have not received alternative GA medications or therapies in the study eye.

For this estimand, data following the below intercurrent event will be dealt with in the following specific way:

Subject receives alternative GA medications or therapies in the study eye: GA lesion size data collected in the study eye after the subject initiates alternative GA medications or therapies will be censored and imputed assuming missing at random.

#### Handling of missing values not related to intercurrent event 2.5.4

For missing data not related to the defined intercurrent event, the estimand based on an MAR approach will be considered specifically for each treatment arm the subjects are assigned.

#### 2.5.5 Sensitivity analyses

Not applicable.

#### 2.5.6 Supplementary analyses

Not applicable.

#### 2.6 Analysis supporting secondary objectives

There are six secondary objectives:

- 1. Evaluate the effect of GT005 on the progression of GA in subjects with GA due to AMD
- 2. Evaluate the safety and tolerability of GT005
- 3. Evaluate the effect of GT005 on retinal anatomical measures
- 4. Evaluate the effect of GT005 on functional measures: BCVA and LLD
- 5. Evaluate the effect of GT005 on visual function: MNRead and FRI
- 6. Evaluate the effect of GT005 on patient-reported outcomes

## 2.6.1 Secondary endpoint(s)

The corresponding secondary endpoints are:

- 1. Change from baseline through Week 96 in GA area as measured by FAF
- 2. Frequency of TEAE through Week 96
- 3. Change in retinal morphology on multimodal imaging through Week 96
- 4.a Change in BCVA ETDRS letters through Week 96
- 4.b Change in LLD in ETDRS letters through Week 96
- 5.a Change in reading performance as assessed by MNRead chart through Week 96
- 5.b Change in FRI index through Week 96
- 6. Change in quality of life measured by VFQ-25 through Week 96

# 2.6.2 Statistical hypothesis, model, and method of analysis

- 1. Change from baseline through Week 96 in GA area as measured by FAF
  - MMRM as described in Section 2.5.2 will be applied to the change from baseline through Week 96 in GA area, with intercurrent event and missing data handled in the same way as for the primary estimand (Sections 2.5.3, 2.5.4).

The estimated least-squares mean (LSM) for the change in GA area, and treatment difference against untreated control, as well as the corresponding 90% confidence interval, will be summarized by visit and treatment group. A line plot for the estimated LSM with 90% CI by visit and treatment group will also be provided.

- 2. Frequency of TEAE through Week 96
  - Summary tables for adverse events of special interest (AESI) will be provided as described in Section 2.7.1.1.
  - Summary tables for treatment-emergent serious AE (TESAE) will be presented as described in Section 2.7.1.
  - Subjects who did not receive treatment due to surgical procedure related AEs will be listed separately by treatment group.
- 3. Change in retinal morphology on multimodal imaging through Week 96
  - The presence of the following retinal morphology will be summarized based on observed data by visit for the number and percentage of subjects in reported categories:
    - i. Junctional zone of GA (Increased FAF, Normal FAF, Not Applicable, Cannot Grade) assessed by FAF.
    - ii. Junctional zone patterns (Atypical, Banded, Diffuse, Focal, Cannot Grade) assessed by FAF.

#### 4.a Change in BCVA in ETDRS letters through Week 96

• Change in BCVA through Week 96 will be estimated among treatment groups via least-squares means from MMRM Model. The model will include the change from baseline in BCVA measured by ETDRS as the dependent variable, BCVA at the baseline as the covariate, assessment visit, treatment group, two interaction terms (assessment visit and treatment group, assessment visit and BCVA at the baseline) as the fixed effect and participant as a random effect. The estimated LSM for the change in BCVA, and treatment difference against untreated control, as well as the corresponding 90% confidence interval, will be summarized by visit and treatment group. A line plot for the estimated LSM with 90% CI by visit and treatment group will also be provided. All BCVA assessments will be listed by treatment group, site, and subject.

## 4.b Change in LLD in ETDRS letters through Week 96

- The LLD and the changes from baseline will be summarized based on observed data by assessment visit and treatment group.
- 5.a Change in reading performance as assessed by MNRead chart through Week 96
  - The Maximum reading speed (MRS) for each eye as assessed by MNRead Chart and change from baseline will be summarized based on observed data by visit and treatment group. Reading speed (words per minute) will be computed for each of the 19 sentences read using the following formula:

 $60 \times max(0,10 - number\ of\ errors)/reading\ time\ in\ seconds$ 

The mean of three higher reading speeds will be reported as the maximum reading speed.

- 5.b Change in FRI index through Week 96
  - The FRI index and the changes from baseline will be calculated and summarized based on observed data by assessment visits and treatment group.
- 6. Change in quality of life measured by VFQ-25 through Week 96
  - The VFQ-25 sub-scales and composite scores and the changes from baseline will be calculated and summarized based on observed data by assessment visits and treatment group.

#### 2.6.3 Handling of missing values/censoring/discontinuations

Missing data handling of secondary endpoints are specified in Section 2.6.2.

### 2.7 Safety analyses

For all safety analyses, the FAS will be used. All listings and tables will be presented by the treatment group.

# 2.7.1 Adverse events (AEs)

Only AEs that occurred during the study period (from the date of randomization to the end of study) will be summarized. AEs recorded after screening but before the date of randomization will be listed only.

**Treatment-emergent Adverse Event** (TEAE): An adverse event is considered treatment emergent if the start date/time of the event is on or after the date of randomization, irrespective of the treatment arm. The primary summaries of AEs will be based on TEAEs.

The number and percentage of subjects with AEs will be summarized separately for ocular (study eye and fellow eye) and non-ocular events by treatment group in the following ways unless otherwise specified:

- Overall summary of death, subjects with any AE, any severe AE, any study treatment-related AE, any surgical procedure related AE, any AE leading to study discontinuation, any serious AE (SAE), any study treatment-related SAE, any surgical procedure related SAE, any SAE leading to study discontinuation
- AEs by primary SOC and PT
- AEs related to study treatment by SOC and PT (separately for study eye and non-ocular)
- AEs related to surgical procedure by SOC and PT (separately for study eye and non-ocular)
- SAEs by primary SOC and PT
- SAEs related to study treatment by SOC and PT (separately for study eye and non-ocular)
- SAEs related to surgical procedure by SOC and PT (separately for study eye and non-ocular)

A subject with multiple adverse events within a primary SOC is only counted once towards the total of the primary SOC.

All AEs, deaths, and SAEs (including those from the pre- and post-treatment periods) will be listed and those collected after the use of alternative GA therapies/medications, or during the pre-treatment, post-study period will be flagged. In addition, subjects who are not receiving treatment due to surgical procedure-related AEs will be listed separately by treatment group.

The MedDRA version used for reporting the AEs will be described in footnote.

For the legal requirements of ClinicalTrials.gov and EudraCT, two required tables on "ontreatment/treatment emergent" adverse events which are not serious adverse events with an incidence greater than 2% (or other cutting point as appropriate) and on "on-treatment/treatment emergent" serious adverse events and SAE suspected to be related to study treatment will be provided by system organ class and preferred term on the safety set population (i.e., the FAS of this study).

If for the same subject, several consecutive AEs (irrespective of study treatment causality, seriousness and severity) occurred with the same SOC and PT:

- a single occurrence will be counted if there is ≤ 1 day gap between the end date of the preceding AE and the start date of the consecutive AE
- more than one occurrence will be counted if there is > 1 day gap between the end date of the preceding AE and the start date of the consecutive AE

For occurrence, the presence of at least one SAE/SAE suspected to be related to study treatment/non-SAE has to be checked in a block e.g., among AEs in a  $\leq$  1 day gap block, if at least one SAE is occurring, then one occurrence is calculated for that SAE.

The number of deaths resulting from SAEs suspected to be related to study treatment and SAEs irrespective of study treatment relationship will be provided by SOC and PT.

# 2.7.1.1 Adverse events of special interest / grouping of AEs

An AESI (serious or non-serious) is one of scientific and medical concern specific to the Sponsor's product or program, for which ongoing monitoring and rapid communication by the Investigator to the Sponsor can be appropriate. AESIs should also be assessed as to whether it fits the criteria of an SAE and reported appropriately. AESI should be reported as per reporting requirements [Protocol Section 8.5.1].



The number and percentage of subjects with AESIs will be summarized separated for ocular (study eye and fellow eye) events by category, PT, and treatment group. In addition, AESIs related to the study treatment and/or surgical procedure will be summarized by category, PT and treatment group.

#### 2.7.2 Deaths

All deaths will be summarized by primary SOC and PT. A listing will also be provided.

#### 2.7.3 Loss in best corrected visual acuity

The number and the percentage of subjects who lost  $\geq 15/\geq 30$  letters in BCVA from baseline up to Week 96 will be presented for the study eye and the fellow eye. Missing data will not be imputed.

Page 22 of 34

#### 2.7.4 Laboratory data

Laboratory parameters listed in Table 2-1 will be presented graphically using boxplots of absolute change from baseline values by treatment group and visit. No summary by visit tables will be provided.

A summary table with number and percentage of subjects satisfying the criteria representing clinically relevant abnormalities defined in Table 2-1 at any visit will be presented. A listing of subjects satisfying at least one criterion in Table 2-1 at any visit will also be presented.

Table 2-1 Clinically notable laboratory values

| Test | Critically Low | Critically High | Units |
|------------------|----------------|-----------------|----------|
| Hemoglobin | < 7.0 | > 20.0 | g/dL |
| White Cell Count | < 2.0 | > 35.0 | x10E3/uL |
| Platelets | < 50 | > 1000 | x10E3/uL |
| Glucose | < 40 | > 500 | mg/dL |
| Calcium | < 6.0 | > 12.0 | mg/dL |
| Phosphate | < 0.9 | | mg/dL |
| Sodium | < 120 | > 160 | mmol/L |
| Potassium | < 3.0 | > 6.0 | mmol/L |
| Magnesium | < 0.74 | > 1.0 | mmol/L |
| AST | | 41 | U/L |
| ALT | | 45 | U/L |
| Total bilirubin | | 21 | umol/L |

#### 2.7.5 Other safety data

#### 2.7.5.1 ECG and cardiac imaging data

No applicable.

### **2.7.5.2** Vital signs

A listing of subjects satisfying at least one criterion in Table 2-2 at any visit will be presented.

Table 2-2 Clinically notable vital signs

| Variable | Category | Critical values |
|---|---|---|
| Systolic blood | High | Either >180 with an increase from baseline >30 or >200 absolute |
| pressure (mmHg) | Low | Either <90 with a decrease from baseline >30 or <75 absolute |
| Diastolic blood | High | Either >105 with an increase from baseline >20 or >115 absolute |
| pressure (mmHg) | Low | Either <50 with a decrease from baseline > 20 or <40 absolute |
| Pulse rate (bpm) | High | Either >120 with an increase from baseline of >25 or > 130 |
| , | _ | absolute |
| | Low | Either <50 with a decrease from baseline >30 or <40 absolute |

# 2.8 Pharmacokinetic endpoints

Not applicable.

# 2.9 PD and PK/PD analyses

Not applicable.

## 2.10 Patient-reported outcomes

# Functional Reading Independence (FRI) Index

The FRI index is a new patient-reported outcome measure developed specifically for use in GA patients. The FRI index evaluates the level of independence patients have in performing everyday activities that require reading, such as writing a cheque or reading a prescription. Scores derived from the index range from 1 (unable to do) to 4 (total independence).

The composite score is the sum of the seven sub-questions.

If responses are missing for main questions or sub-questions, scores may be imputed based on the scoring for missing items algorithm provided in Table 2-3 below.

Table 2-3 Scoring missing FRI items

| Question or sub-question with | Missing response within context of other | Coding and imputation |
|---|---|---|
| missing data | sub-questions | |
| | If missing main question and responses of "Yes" or "No" to sub-questions a-e | Impute "Yes" to main question and score according to algorithm |
| Main Questions 1–7 | If missing main question and "Your vision" or "For other reasons" to sub-question g | Impute "No" to main question and score according to algorithm |
| | If missing main question and no responses to any subquestions | Code as "missing" |
| Sub-questions a–c | If missing sub-questions a-c | Code as "missing" and score according to algorithm |
| Sub-question d | If missing sub-question d and "No" response to all sub-<br>questions a-c | Impute "No" for sub-question d and score according to algorithm |
| Sub question a | If "Yes" to performing activity<br>and "missing" for sub-question<br>e and no responses to sub-<br>question f | Impute "No" for sub-question e and score according to algorithm |
| Sub-question e | If "Yes" to performing activity<br>and "missing" for sub-question<br>e and response of "Some of the<br>time", "Most of the time" or | Impute "yes" for sub-question e and score according to algorithm |

| COI | IIIQ | eni | lai |
|-----|------|-----|-----|

| | "All of the time" to subquestion f | |
|---|---|---|
| Sub-question f | If "Yes" to performing activity, "Yes" to sub-question e and "missing" for sub-question f | Impute "Some of the time" for sub-question f and score according to algorithm |
| Sub-question g | If "No" to main question and "missing" for sub-question g | Impute "For other reasons" for<br>sub-question g and score<br>according to algorithm |

#### **Visual Function Questionnaires (VFQ-25)**

The VFQ-25 consists of a base set of 25 vision-targeted questions representing 11 vision-related constructs, plus an additional single-item general health rating question. The VFQ-25 subscales and composite scores and changes from baseline will be calculated and summarized by assessment visit. Each subscale score has a range of 0 to 100 inclusive and will be calculated from the re-scaled raw data as described in Table 2-4. A missing response will not be re-scaled (except for the response to question 15c, see below, which will be re-set to 0 if the response to question 15b is 1).

Table 2-4 **Rescaling of VFQ-25 questions** 

| Answer to question | Rescaling for<br>questions 1, 3, 4<br>and 15c | Rescaling for question 2 | Rescaling for questions 5-14, 16 and 16a | Rescaling for questions 17-25 |
|---|---|---|---|---|
| 1 | 100 | 100 | 100 | 0 |
| 2 | 75 | 80 | 75 | 25 |
| 3 | 50 | 60 | 50 | 50 |
| 4 | 25 | 40 | 25 | 75 |
| 5 | 0 | 20 | 0 | 100 |
| 6 | N/A | 0 | N/A* | N/A |

Item 15c has four-response levels, but is expanded to a five-levels using item 15b.

Note: If 15b=1, then 15c should be recoded to "0"

If 15b=2, then 15c should be recoded to missing

If 15b=3, then 15c should be recoded to missing

The subscale scores are then calculated according to Table 2-5.

Table 2-5 Questions contributing to VFQ-25 subscales

| Subscale | Questions |
|---------------------|------------------|
| General vision | 2 |
| Ocular pain | 4 and 19 |
| Near activities | 5, 6 and 7 |
| Distance activities | 8, 9 and 14 |
| Social functioning | 11 and 13 |
| Mental health | 3, 21, 22 and 25 |
| Role difficulties | 17 and 18 |

<sup>\*</sup>Response choice "6" indicates that the person does not perform the activity because of non-vision related problems. If this choice is selected, the item is coded as "missing".

| Novartis | Confidential | Page 25 of 34 |
|-----------------|--------------|-------------------------|
| SAP Amendment 3 | | Study No. CPPY988A12201 |

| Dependency | 20, 23 and 24 |
|-------------------|-----------------|
| Driving | 15c, 16 and 16a |
| Color vision | 12 |
| Peripheral vision | 10 |

The composite score is the average of the 11 subscales shown in Table 2-5. It will be set to missing if at least six of the subscales are missing.







# 2.13 Data analysis at Week 48

The Week 48 analysis will be performed when all subjects completed the Week 48 visit or terminated the study prior to Week 48. The objective of this analysis is to demonstrate the effect of GT005 vs untreated control on the progression of GA in subjects with GA due to AMD. The following analyses will be presented:

- Subject disposition, demographics at baseline, and ocular baseline characteristics
- Concurrent procedures
- Subject exposure and treatment compliance
- Analysis corresponding to the primary objective, as described in Section 2.5
- Analyses corresponding to secondary objectives:
  - To evaluate the safety and tolerability of GT005
  - o To evaluate the effect of GT005 on functional measures
- Summary tables of the following AE/SAE and AESI with onset date prior to/on the cut-off date of the Week 48 analysis will be generated separately for ocular (study eye and fellow eye) and non-ocular events by treatment and in total:
  - Overall summary of subjects with death, any AE, any severe AE, any study treatment-related AE, any surgical procedure related AE, any AE leading to study discontinuation, any serious SAE, any study treatment-related SAE, any surgical procedure related SAE, any SAE leading to study discontinuation
  - AEs by primary SOC and PT
  - AEs related to study treatment by SOC and PT (only for study eye and nonocular)

- AEs related to surgical procedure by SOC and PT (only for study eye and non-ocular)
- SAEs by primary SOC and PT
- o SAEs related to study treatment by SOC and PT (only for study eye)
- SAEs related to surgical procedure by SOC and PT (only for study eye and non-ocular)
- Ocular AESI by category
- Deaths will be summarized by SOC and PT by treatment arm and in total

# 3 Sample size calculation

Untreated control mean GA change at 72 weeks was assumed to be 3.0 mm<sup>2</sup> with standard deviation (SD) =1.5 mm<sup>2</sup>. The following hypotheses are considered:

$$\begin{split} H0_M: \; \mu_M - \mu_C &= 0, \; HA_M: \; \mu_M - \mu_C < 0 \\ H0_H: \; \mu_H - \mu_C &= 0, \; HA_H: \; \mu_H - \mu_C < 0 \end{split}$$

Where  $\mu_M$ ,  $\mu_H$  and  $\mu_C$  represent the unknown true mean GA change on FAF at 72 weeks in the GT005 medium dose [1005], GT005 high dose [1006], and pooled untreated control, respectively.

The total sample size planned is approximately 250, accounting for an estimated 15% of subjects that are expected to discontinue treatment and not provide the target 72-week observation; hence power calculations are based on n=70 per treatment group (GT005 medium dose GT005 high dose pooled untreated control).



# 4 Change to protocol specified analyses

| A single | interim a | analysis | for futility | will | be | performed | when | approximately | 60% | of subj | jects |
|---|---|---|---|---|---|---|---|---|---|---|---|
| have GA | data ava | ilable at | Week 48. | | | | | | | | |



The Safety Analysis Set (SAF) was removed.

A Week 48 analysis was added as an interim analysis and the primary endpoint at Week 72 will be performed during the final CSR.

# 5 Appendix

Statistical methods are described in the main part of the clinical study report. This appendix provides further details on missing data imputation, statistical methods, and statistical derivation.

## 5.1 Imputation rules

The general approach to handling missing dates is shown below for dates of AEs, medical history diagnosis, and concomitant treatment. The imputation of missing dates for surgery or procedures will use the same rules as for concomitant treatment.

The detailed algorithms will appear in Programming Dataset Specifications.

For the purpose of date imputation, the treatment follow-up period date is defined as the last available visit date.

### 5.1.1 AE date imputation

#### 5.1.1.1 Adverse event end date imputation

- 1. If the AE end date month is missing, the imputed end date should be set to the earliest of the (treatment follow up period date, 31DECYYYY, date of death, cut-off date if available).
- 2. If the AE end date day is missing, the imputed end date should be set to the earliest of the (the last visit date, last day of the month, date of death, cut-off date if available).
- 3. If AE year is missing or AE is ongoing, the end date will not be imputed.
- 4. In case the imputed AE end date is before AE start date, then use AE start date as imputed AE end date.

#### 5.1.1.2 Adverse event start date imputation

The following table explains the notation used in the logic matrix. Please note that **missing** start dates will not be imputed.

| | Day | Month | Year |
|-------------------------------------|----------|-------|-------|
| Partial Adverse Event<br>Start Date | Not used | MON | YYYY |
| Randomization Date | Not used | RANDM | RANDY |

The following matrix explains the logic behind the imputation.

| | MON<br>MISSING | MON < RANDM | MON = RANDM | MON > RANDM |
|---|---|---|---|---|
| YYYY | (1) | (1) | (1) | (1) |
| MISSING | No convention | No convention | No convention | No convention |
| YYYY < TRTY | ( 2.a ) | ( 2.b ) | ( 2.b ) | ( 2.b ) |
| | Before Randomization | Before Randomization | Before Randomization | Before Randomization |
| YYYY = TRTY | ( 4.a ) | ( 4.b ) | ( 4.c ) | ( 4.c ) |
| | Uncertain | Before Randomization | Uncertain | After Randomization |
| YYYY > TRTY | ( 3.a ) | ( 3.b ) | ( 3.b ) | ( 3.b ) |
| | After Randomization | After Randomization | After Randomization | After Randomization |

Before imputing AE start date, find the AE start reference date.

- 1. If the (imputed) AE end date is complete and the (imputed) AE end date < randomization date then AE start reference date = min (informed consent date, earliest visit date).
- 2. Else AE start reference date = randomization date

## Impute AE start date -

- 1. If the AE start date year value is missing, the date uncertainty is too high to impute a rational date. Therefore, if the AE year value is missing, the imputed AE start date is set to NULL.
- 2. If the AE start date year value is less than the randomization date year value, the AE started before randomization. Therefore:
  - a. If AE day and month are missing, the imputed AE start date is set to the mid-year point (01JulYYYY).
  - b. If AE month is missing but day is not missing, the observed start date will be used with month imputed as JulYYYY.
  - c. Else if AE month is not missing, the imputed AE start date is set to the midmonth point (15MONYYYY).
- 3. If the AE start date year value is greater than the randomization date year value, the AE started after randomization. Therefore:
  - a. If the AE day and month are missing, the imputed AE start date is set to the year start point (01JanYYYY).
  - b. If AE month is missing but day is not missing, the observed start date will be used with month imputed as JulYYYY.
  - c. Else if the AE month is not missing, the imputed AE start date is set to the later of (month start point (01MONYYYY), AE start reference date + 1 day).
- 4. If the AE start date year value is equal to the randomization date year value:
  - a. And the AE day and month are missing the imputed AE start date is set to the AE reference start date + 1 day.
  - b. If AE month is missing and day is not missing, the observed start date will be used with month imputed as the reference start month.
  - c. Else if the AE month is less than the randomization month, the imputed AE start date is set to the mid-month point (15MONYYYY).
  - d. Else if the AE month is equal to the randomization date month or greater than the randomization date month, the imputed AE start date is set to the later of (month start point (01MONYYYY), AE start reference date + 1 day).

If complete (imputed) AE end date is available and the imputed AE start date is greater than the (imputed) AE end date, then imputed AE start date should be set to the (imputed) AE end date.

#### 5.1.2 **Concomitant medication date imputation**

#### 5.1.2.1 Concomitant treatment end date imputation

- 1. If CM end day is missing and CM month/year are non-missing then impute CM day as the minimum of the last study visit date and the last day of the month.
- 2. If CM end day/month are missing and CM year is non-missing then impute CM day as the minimum of the last study visit date and the end of the year (31DECYYYY).
- 3. Only include if ongoing records will have an imputed CM end date. If CM day/month/year is missing then use the last study visit date + 1 day as the imputed CM end date.
- 4. If imputed CM end date is less than the CM start date, use the CM start date as the imputed CM end date.
- 5. If imputed CM end date is greater than date of death, date of cutoff, or the last visit date, then use the minimum of date of death, date of cutoff, and the last visit date as the imputed CM end date.

### 5.1.2.2 Concomitant treatment start date imputation

The following table explains the notation used in the logic matrix. Please note that missing start dates will not be imputed.

| | Day | Month | Year |
|------------------------|----------|-------|-------|
| Partial CMD Start Date | Not used | MON | YYYY |
| Randomization Date | Not used | RANDM | RANDY |

The following matrix explains the logic behind the imputation.

| C | MON<br>MISSING | MON < RANDM | MON = RANDM | MON > RANDM |
|---|---|---|---|---|
| YYYY | (1) | (1) | (1) | (1) |
| MISSING | Uncertain | Uncertain | Uncertain | Uncertain |
| YYYY < TRTY | ( 2.a ) | ( 2.b ) | ( 2.b ) | ( 2.b ) |
| | Before Randomization | Before Randomization | Before Randomization | Before Randomization |
| YYYY = TRTY | ( 4.a ) | (4.b) | ( 4.a ) | ( 4.c ) |
| | Uncertain | Before Randomization | Uncertain | After Randomization |
| YYYY > TRTY | ( 3.a ) | (3.b) | (3.b) | ( 3.b ) |
| | After Randomization | After Randomization | After Randomization | After Randomization |

If the CM start date year value is missing, the imputed CM start date is set to one day prior to randomization date.

If the CM start date year value is less than the randomization date year value, the CM started before randomization. Therefore:

a. If the CM day and month are missing, the imputed CM start date is set to the mid-year point (01JulYYYY).

- b. If CM month is missing but day is not missing, the observed start date will be used with month imputed as JulYYYY.
- c. Else if the CM month is not missing, the imputed CM start date is set to the mid-month point (15MONYYYY).

If the CM start date year value is greater than the randomization date year value, the CM started after randomization. Therefore:

- a. If the CM day and month are missing, the imputed CM start date is set to the year start point (01JanYYYY).
- b. If CM month is missing but day is not missing, the observed start date will be used with month imputed as JanYYYY.
- c. Else if the CM month is not missing, the imputed CM start date is set to the month start point (01MONYYYY).

If the CM start date year value is equal to the randomization date year value:

- a. And the CM day and CM month are missing or the CM day is missing and CM month is equal to the randomization date month, then the imputed CM start date is set to one day prior randomization date.
- b. Else if the CM month is less than the randomization date month, the imputed CM start date is set to the mid-month point (15MONYYYY).
- c. Else if the CM month is greater than the randomization date month, the imputed CM start date is set to the month start point (01MONYYYY).

If complete (imputed) CM end date is available and the imputed CM start date is greater than the (imputed) CM end date, then imputed CM start date should be set to the (imputed) CM end date.

## 5.1.2.3 Medical history date of diagnosis imputation

Completely missing dates and partially missing end dates will not be imputed. Partial dates of diagnosis will be compared to the randomization date.

- If DIAG year < randomization date year and DIAG month is missing, the imputed DIAG date is set to the mid-year point (01JULYYYY)
  - else if DIAG month is not missing, the imputed DIAG date is set to the mid-month point (15MONYYYY)
- If DIAG year = randomization date year
  - and (DIAG month is missing OR DIAG month is equal to randomization month), the imputed DIAG date is set to one day before randomization date
  - else if DIAG month < randomization month, the imputed DIAG date is set to the midmonth point (15MON YYYY)
  - else if DIAG month > randomization month => data error
- If DIAG year > randomization date year => data error

#### 5.1.2.4 Other imputations

Not applicable.

# 5.2 AEs coding/grading

Adverse events are coded using the Medical Dictionary for Regulatory Activities (MedDRA) terminology.

The below severity grade will be used in this study:

- Mild: usually transient in nature and generally not interfering with normal activities
- Moderate: sufficiently discomforting to interfere with normal activities
- Severe: prevents normal activities

## 5.3 Laboratory parameters derivations

Not applicable.

### 5.4 Statistical models

#### 5.4.1 Analysis supporting primary objective(s)

The following MMRM will be used for the primary efficacy endpoint. The model will include the change from baseline in GA area measured by FAF as the dependent variable, GA area at the baseline as the covariate, assessment visit, treatment group, two interaction terms (assessment visit and treatment group, assessment visit and GA area at the baseline) as the fixed effect and participant as a random effect.

For this analysis, the data structure is one record per subject per scheduled visit. The data will include all subjects and have records for all scheduled visits, regardless of whether the assessment was missed or not at a given visit. Missing values will not be imputed and will be passed to the model as missing. The SAS PROC MIXED will be used to perform the analysis.

### 5.5 Rule of exclusion criteria of analysis sets

The below classification of non-PDs will be used for the analysis sets.

Table 5-1 Subject Classification

| Analysis Set | Non-PD criteria that cause participants to be excluded |
|-------------------|--------------------------------------------------------|
| All Enrolled Set | Not signed the informed consent |
| Full Analysis Set | Not randomized |

# 6 References

Bretz, F. a. (2017). Multiple test strategies for comparing several doses with a control in confirmatory trials from Handbook of Methods for Designing, Monitoring, and Analyzing Dose-Finding Trials. Chapman and Hall/CRC.